CLINICAL TRIAL: NCT04815954
Title: Early vs Late Urinary Catheter Removal After Renal Transplantation Randomised Clinical Trial
Brief Title: Early vs Late Urinary Catheter Removal After Renal Transplantation
Acronym: ELUCATR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, PAWEŁ STUDNICKI, Principal Investigator, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Not assigned
Record Dates: First submitted 2020-02-10; First posted 2021-03-25 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Kidney Transplant; Complications; Kidney Transplant Infection; Urinary Fistula; Urinary Tract Infections; Urinary Catheter
Keywords: kidney transplant; urinary tract infections; foley catheter; urinary catheter; urinary fistula; urethral stricture
MeSH Terms: conditions — Urinary Fistula; Urinary Tract Infections; Urethral Stricture

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: Randomisation will be supervised centrally by the leader center. Generated numbers will be closed in non-transparent envelopes numbered sequentially and shipped to each participating center. A center is supposed to use the envelopes for group assignment consecutively with increasing numbers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early group (Experimental): Early urinary catheter removal: 24±6 hours after completion of surgery.
  Interventions: Procedure: Urinary catheter removal
- Delayed group (Active Comparator): Delayed urinary catheter removal: 72±6 hours after completion of surgery.
  Interventions: Procedure: Urinary catheter removal

INTERVENTIONS:
Procedure: Urinary catheter removal — Removal of urinary catheter which was placed during kidney transplantation.

SUMMARY:
The purpose of this study is to compare frequency of UTI, urine leak and need for reoperation in patients after renal transplant with early or delayed Foley catheter removal. The hypothesis of the ELUCATR trial is that there is no need to keep Foley catheter longer than 24 hours after kidney transplant due to lack of significant effect on urological complications (urine leak, ureter strictures). Early removal can also reduce urinary tract infections.

Main advantage of urinary catheter placement is continual diuresis monitoring and lower bladder pressure. Some hypothesize that increased pressure can disrupt ureteroneocystostomy with resultant urinary fistula. Clinical practice is to remove the catheter between 1-10 post-transplant day. Only few studies described removal of Foley catheter in the first 48 hours. There is no level 1 evidence for timing of urinary catheter removal after kidney transplantation.

Urinary tract infection is a common complication after KTx occurring in about 7-80% patients. Studies suggest direct negative effect of UTI on long-term renal allograft function. There are several independent risk factors for developing UTI: female sex, diabetes and obesity. Duration of catheterization is a modifiable risk factor.

Urine leak and ureter stenosis are relatively frequent surgical complications of kidney transplantation. Urine leaks occur in 2-9% of all kidney transplants. Most of them happen within 3 months after surgery. Urinary fistula contributes to mortality and graft loss. Majority of them need intervention with nephrostomy, pigtail ureteral stent or surgery. Anastomotic or ureter stenosis occurs in 3.1% of all kidney transplants and is usually resolved with open ureteroneocystostomy. Diagnosed and treated early, it does not affect patient and graft survival. There are no solid data documenting influence of the urinary bladder catheterization on fistulas, urinomas, ureter strictures and need for reoperation in this set of patients.

European Best Renal Practice Guidelines recommend removal of the catheter as early as possible, however a randomized trial on timing and adverse event rates (urinary tract infection, urinary leakage) is needed.

DETAILED DESCRIPTION:
1. Objectives of the study

   1. Main aim of the study:

      Early urinary catheter removal is safe and does not increase urinary complications rate. Zero hypothesis is that early and delayed Foley catheter removal have similar urinary complications rate (urinary fistula, urinary tract infections). Alternative hypothesis is that early catheter removal decreases urinary tract infections.
   2. Primary endpoints:

      * Urinary fistula or stenosis requiring intervention,
      * 30 day graft function measured as serum creatinine,
      * 1 year graft survival and function.
   3. Secondary endpoints:

      * Urinary tract infections,
      * BK virus infection,
      * length of hospital stay.
2. Patients and Methods

2.1 Study organisation

The study has been designed as a randomized, controlled, open label, multicenter trial to compare urinary complications rate between early and delayed Foley catheter removal groups in kidney transplant recipients. Computer list of random numbers will be generated, even numbers will be assigned to early and odd numbers to late catheter removal, 1:1 randomisation ratio is expected. At least 3 large-volume renal transplant centers will participate in the study. Randomisation will be supervised centrally by the leader center. Generated numbers will be closed in non-transparent envelopes numbered sequentially and shipped to each participating center. A center is supposed to use the envelopes for group assignment consecutively with increasing numbers. A record of computer-generated number and envelope number will be stored at the leader center. An institutional review board of the Medical University of Warsaw accepted the study design and patient information leaflet. MS Access-based electronic case report file will be used. CRFs will be checked for completeness and concordance with source documents and adherence to the study protocol by the study leader.

2.2 Study design

Donor and pre-transplant recipient data will be noted in a database. Donor blood, urine and preservation solution will be cultured, 10^5 colonies in the former is considered significant. Important transplant anatomical features, like multiple renal arteries will be noted. After screening and informed consent of the patient for participation in the study, kidney transplantation will be performed. Single dose of cefazolin adjusted for patient weight will be administered 30 minutes prior to skin incision. Other options of antibiotic prophylaxis or preemptive treatment are acceptable, however agent and duration must be noted in an electronic Case Report File (CRF). At the beginning of surgical procedure in the operating room, sterile catheterization of the urinary bladder and microbiology sampling will be performed. After uneventful vascular anastomosis, neoureterocystostomy will be done with Lich-Gregoire or a variation of U-stitch technique (McKinnon, other typical). Ureteral stent will be placed at surgeon's discretion. Suction drainage will be positioned in graft proximity. After wound closure and completion of the surgery, inclusion and exclusion criteria will be evaluated. Intraoperative data (blood loss, surgery duration, cold ischemia time, details of the anastomosis, utilization of magnifying loupes, pigtail placement) will be noted.

2.3 Eligibility and exclusion criteria.

2.3.1 Inclusion criteria

* Age>18
* Kidney transplant recipient
* Informed consent signed

2.3.2 Exclusion criteria BMI<18 or >40 kg/m2 Significant anatomical abnormalities of lower urinary tract Previous surgery on bladder or urinary tract Unusual urinary anastomosis (Leadbetter-Politano, Boari, conduit, psoas hitch, pyelo-ureteral or uretero-ureteral, double ureter) Severe vascular complications during surgery with blood loss >1000 ml Haemodynamic shock or profund instability after surgery

Participants will be randomised to a group early urinary catheter removal (EG) or delayed removal group (DG). Early catheter removal will be done 24±6 hours after surgery. In a delayed group catheter will be removed 72±6 hours after completion of surgery. Shorter or longer catheterization will be considered protocol violation and reasons for ought to be explained in source documents and CRF.

Suction drain will be removed when discharge volume falls below 50 ml/day. If clear discharge (>100 ml/day) continues for 2 consecutive days, discharge fluid and serum creatinine ought to be measured. If fluid creatinine exceeds its serum concentration by at least 30%, urine leakage will be diagnosed and appropriate intervention applied according to surgeon's clinical judgement. Only fistulas requiring medical intervention: reintroduction of the catheter, endoscopic stenting, nephrostomy or surgery will be considered significant and fulfill criteria for primary endpoint of the study.

The course of study will consist of screen visit, hospitalization (with the transplantation procedure, catheter removal, follow up after 48h after catheter removal), follow up visit at 15 days after procedure and follow up visit at 30 days after procedure (see table 2). Patients with urinary complications (fistula, stenosis, infection) will have additional visits every 30 days until complete resolution of complication. Patients with stented anastomosis who will not have a pigtail removed until day 30 will be followed till 7 days after stent removal or resolution of complications would any occur. A final visit 1 year after transplantation will assess patient and graft survival, kidney function, late urinary complications beyond one month from transplantation.

2.4 Sample size and statistics

The investigators assumed early catheter removal reduces the risk of UTI by 10% (RR=0.9) and risk of urinary anastomosis complications is comparable. To achieve a power of 80% at p=0,05 an expected sample size is 450 patients divided fairly into 2 groups. An intent-to-treat analysis will be performed. Graft survival analysis and length of hospital stay will be calculated with log-rank test. Renal function will be analysed with Student t test, provided normal distribution of serum creatinine is observed. Chi2 will be used for analysis of urinary complications. Post hoc analysis of donor and recipient entry data will confirm groups being comparable fo UTI and urinary fistula risk factors.

Subgroup analysis in groups with and without urinary stent will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipient
* Informed consent signed

Exclusion Criteria:

* BMI under 18kg/m2
* BMI over 40 kg/m2
* Significant anatomical abnormalities of lower urinary tract
* Previous surgery on bladder or urinary tract
* Unusual urinary anastomosis (Leadbetter-Politano, Boari, conduit, psoas hitch, pyelo-ureteral or uretero-ureteral, double ureter)
* Severe vascular complications during surgery with blood loss >1000 ml
* Underwent haemodynamic shock or profund instability after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2026-03-26 (Estimated); Study Completion 2027-04-26 (Estimated)

PRIMARY OUTCOMES:
Urinary fistula | 1 year
  Presence of urine in the drains or peri-transplant fluid collection demonstrated with biochemical analysis (creatinine in mg/dl in the drains or aspirate exceeding that of serum in mg/dl by at least 30%); symptoms may be present in the first week after transplantation as increased drainage discharge, impaired graft function and decreased diuresis, fluid collection seen in ultrasound, CT or scintigraphy, discharge onto the skin, abdominal pain, cutaneous oedema often towards the scrotum, pain and inflammatory appearance of the scar; volume of the discharge has no influence on diagnosis. Only fistulas requiring medical intervention as reintroduction of the catheter, endoscopic stenting, nephrostomy or surgery will be considered in the study.
Urinary stenosis | 1 year
  Obstruction of the urine outflow from the transplanted kidney causing pelvicalyceal dilatation and impaired graft function; dilatation may be minimal due to fibrosis of the renal tissue and ex juvantibus diagnosis in these cases is acceptable. Only strictures requiring medical intervention as reintroduction of the catheter, endoscopic stenting, nephrostomy or surgery will be considered in the study.
30 day graft function measured as serum creatinine | 30 days
  Serum creatinine in mg/dl
1 year graft survival in days and function measured as serum creatinine | 1 year
  Graft survival in days; serum creatinine in mg/dl

SECONDARY OUTCOMES:
Urinary tract infections | 1 year
  1. asymptomatic bacteriuria defined by the presence of >10^5 bacterial colony forming units per milliliter (CFU/mL) of urine on urine culture with no local or systemic symptoms of UTI,
  2. simple cystitis with the presence of >10^5 CFU/mL on urine culture with local urinary symptoms, such as dysuria, frequency, or urgency, but no systemic symptoms, such as fever or allograft pain,
  3. complicated UTI with the presence of >10^5 CFU/mL on urine culture with fever and allograft pain, chills, malaise or bacteremia with the same organism in urine, or biopsy with findings consistent with pyelonephritis,
  4. recurrent UTI with three or more episodes of UTI in one year
BK virus infection | 1 year
  Diagnosed with histopathology and positive immunohistochemistry staining for BK SV40 T antigen; in highly suspicious clinical cases prolonged (>2 weeks) urinary viral shedding with significant BK load (>10 000 copies/ mL) as presumptive diagnosis is also acceptable.
Length of hospital stay | 1 year
  Length of hispital stay in days.

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Studnicki, MD, Principal Investigator — Department of General and Transplantation Surgery, Medical University of Warsaw
Locations (1):
- Department of General and Transplantation Surgery, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brar S, Wang Y, Cannitelli A, Lambadaris M, Li Y, Famure O, Husain S, Kim SJ. Bacteremia in kidney transplant recipients: Burden, causes, and consequences. Clin Transplant. 2019 Mar;33(3):e13479. doi: 10.1111/ctr.13479. Epub 2019 Feb 8. PMID 30650217
- [Background] Goldman JD, Julian K. Urinary tract infections in solid organ transplant recipients: Guidelines from the American Society of Transplantation Infectious Diseases Community of Practice. Clin Transplant. 2019 Sep;33(9):e13507. doi: 10.1111/ctr.13507. Epub 2019 Mar 28. PMID 30793386
- [Background] Akbari R, Rahmani Firouzi S, Akbarzadeh-Pasha A. Old habits die hard; does early urinary catheter removal affect kidney size, bacteriuria and UTI after renal transplantation? J Renal Inj Prev. 2016 Nov 20;6(1):43-48. doi: 10.15171/jrip.2017.08. eCollection 2017. PMID 28487871
- [Background] Cole T, Hakim J, Shapiro R, Kayler LK. Early urethral (Foley) catheter removal positively affects length of stay after renal transplantation. Transplantation. 2007 Apr 15;83(7):995-6. doi: 10.1097/01.tp.0000259723.92943.8f. No abstract available. PMID 17460573
- [Background] Chuang P, Parikh CR, Langone A. Urinary tract infections after renal transplantation: a retrospective review at two US transplant centers. Clin Transplant. 2005 Apr;19(2):230-5. doi: 10.1111/j.1399-0012.2005.00327.x. PMID 15740560
- [Background] Lempinen M, Stenman J, Kyllonen L, Salmela K. Surgical complications following 1670 consecutive adult renal transplantations: A single center study. Scand J Surg. 2015 Dec;104(4):254-9. doi: 10.1177/1457496914565419. Epub 2015 Jan 7. PMID 25567856
- [Background] Siskind E, Sameyah E, Goncharuk E, Olsen EM, Feldman J, Giovinazzo K, Blum M, Tyrell R, Evans C, Kuncewitch M, Alexander M, Israel E, Bhaskaran M, Calderon K, Jhaveri KD, Sachdeva M, Bellucci A, Mattana J, Fishbane S, D'Agostino C, Coppa G, Molmenti E. Removal of foley catheters in live donor kidney transplant recipients on postoperative day 1 does not increase the incidence of urine leaks. Int J Angiol. 2013 Mar;22(1):45-8. doi: 10.1055/s-0033-1333870. PMID 24436583
- [Background] Abramowicz D, Cochat P, Claas FH, Heemann U, Pascual J, Dudley C, Harden P, Hourmant M, Maggiore U, Salvadori M, Spasovski G, Squifflet JP, Steiger J, Torres A, Viklicky O, Zeier M, Vanholder R, Van Biesen W, Nagler E. European Renal Best Practice Guideline on kidney donor and recipient evaluation and perioperative care. Nephrol Dial Transplant. 2015 Nov;30(11):1790-7. doi: 10.1093/ndt/gfu216. Epub 2014 Jul 9. PMID 25007790
- [Background] Menegueti MG, Pereira MF, Bellissimo-Rodrigues F, Garcia TM, Saber LT, Nardim ME, Muglia VA, Neto MM, Romao EA. Study of the risk factors related to acquisition of urinary tract infections in patients submitted to renal transplant. Rev Soc Bras Med Trop. 2015 May-Jun;48(3):285-90. doi: 10.1590/0037-8682-0098-2015. PMID 26108006
- [Background] Rubin RH. Infectious disease complications of renal transplantation. Kidney Int. 1993 Jul;44(1):221-36. doi: 10.1038/ki.1993.234. No abstract available. PMID 8394951
- [Background] Wilson CH, Rix DA, Manas DM. Routine intraoperative ureteric stenting for kidney transplant recipients. Cochrane Database Syst Rev. 2013 Jun 17;(6):CD004925. doi: 10.1002/14651858.CD004925.pub3. PMID 23771708
- [Background] de Souza RM, Olsburgh J. Urinary tract infection in the renal transplant patient. Nat Clin Pract Nephrol. 2008 May;4(5):252-64. doi: 10.1038/ncpneph0781. Epub 2008 Mar 11. PMID 18334970
- [Background] Ariza-Heredia EJ, Beam EN, Lesnick TG, Cosio FG, Kremers WK, Razonable RR. Impact of urinary tract infection on allograft function after kidney transplantation. Clin Transplant. 2014 Jun;28(6):683-90. doi: 10.1111/ctr.12366. Epub 2014 Apr 27. PMID 24654771
- [Background] Adamska Z, Karczewski M, Cichanska L, Wieckowska B, Malkiewicz T, Mahadea D, Stronka M. Bacterial Infections in Renal Transplant Recipients. Transplant Proc. 2015 Jul-Aug;47(6):1808-12. doi: 10.1016/j.transproceed.2015.03.046. PMID 26293055
- [Background] Ak O, Yildirim M, Kucuk HF, Gencer S, Demir T. Infections in renal transplant patients: risk factors and infectious agents. Transplant Proc. 2013 Apr;45(3):944-8. doi: 10.1016/j.transproceed.2013.02.080. PMID 23622594
- [Background] Saemann M, Horl WH. Urinary tract infection in renal transplant recipients. Eur J Clin Invest. 2008 Oct;38 Suppl 2:58-65. doi: 10.1111/j.1365-2362.2008.02014.x. PMID 18826483
- [Background] Kawecki D, Wszola M, Kwiatkowski A, Sawicka-Grzelak A, Durlik M, Paczek L, Mlynarczyk G, Chmura A. Bacterial and fungal infections in the early post-transplant period after kidney transplantation: etiological agents and their susceptibility. Transplant Proc. 2014 Oct;46(8):2733-7. doi: 10.1016/j.transproceed.2014.09.115. PMID 25380905
- [Background] Rabkin DG, Stifelman MD, Birkhoff J, Richardson KA, Cohen D, Nowygrod R, Benvenisty AI, Hardy MA. Early catheter removal decreases incidence of urinary tract infections in renal transplant recipients. Transplant Proc. 1998 Dec;30(8):4314-6. doi: 10.1016/s0041-1345(98)01423-7. No abstract available. PMID 9865370
- [Background] Ariza-Heredia EJ, Beam EN, Lesnick TG, Kremers WK, Cosio FG, Razonable RR. Urinary tract infections in kidney transplant recipients: role of gender, urologic abnormalities, and antimicrobial prophylaxis. Ann Transplant. 2013 May 6;18:195-204. doi: 10.12659/AOT.883901. PMID 23792521
- [Background] Guler S, Cimen S, Hurton S, Molinari M. Risks and Benefits of Early Catheter Removal After Renal Transplantation. Transplant Proc. 2015 Dec;47(10):2855-9. doi: 10.1016/j.transproceed.2015.10.032. PMID 26707302
- [Background] Karakayali H, Emiroglu R, Arslan G, Bilgin N, Haberal M. Major infectious complications after kidney transplantation. Transplant Proc. 2001 Feb-Mar;33(1-2):1816-7. doi: 10.1016/s0041-1345(00)02694-4. No abstract available. PMID 11267526
- [Background] Pelle G, Vimont S, Levy PP, Hertig A, Ouali N, Chassin C, Arlet G, Rondeau E, Vandewalle A. Acute pyelonephritis represents a risk factor impairing long-term kidney graft function. Am J Transplant. 2007 Apr;7(4):899-907. doi: 10.1111/j.1600-6143.2006.01700.x. Epub 2007 Feb 7. PMID 17286620
- [Background] Mohan MVNLR, Neeraja M, Sudhaharan S, Raju SB, Gangadhar T, Lakshmi V. Risk Factors for Urinary Tract Infections in Renal Allograft Recipients: Experience of a Tertiary Care Center in Hyderabad, South India. Indian J Nephrol. 2017 Sep-Oct;27(5):372-376. doi: 10.4103/ijn.IJN_331_16. PMID 28904433
- [Background] Tissot E, Limat S, Cornette C, Capellier G. Risk factors for catheter-associated bacteriuria in a medical intensive care unit. Eur J Clin Microbiol Infect Dis. 2001 Apr;20(4):260-2. doi: 10.1007/s100960100480. PMID 11399016
- [Background] Letica-Kriegel AS, Salmasian H, Vawdrey DK, Youngerman BE, Green RA, Furuya EY, Calfee DP, Perotte R. Identifying the risk factors for catheter-associated urinary tract infections: a large cross-sectional study of six hospitals. BMJ Open. 2019 Feb 21;9(2):e022137. doi: 10.1136/bmjopen-2018-022137. PMID 30796114
- [Background] Meddings J, Saint S. Disrupting the life cycle of the urinary catheter. Clin Infect Dis. 2011 Jun;52(11):1291-3. doi: 10.1093/cid/cir195. No abstract available. PMID 21596672
- [Background] Chenoweth C, Saint S. Preventing catheter-associated urinary tract infections in the intensive care unit. Crit Care Clin. 2013 Jan;29(1):19-32. doi: 10.1016/j.ccc.2012.10.005. PMID 23182525
- [Background] Shuman EK, Chenoweth CE. Urinary Catheter-Associated Infections. Infect Dis Clin North Am. 2018 Dec;32(4):885-897. doi: 10.1016/j.idc.2018.07.002. Epub 2018 Sep 18. PMID 30241712
- [Background] Hooton TM, Bradley SF, Cardenas DD, Colgan R, Geerlings SE, Rice JC, Saint S, Schaeffer AJ, Tambayh PA, Tenke P, Nicolle LE; Infectious Diseases Society of America. Diagnosis, prevention, and treatment of catheter-associated urinary tract infection in adults: 2009 International Clinical Practice Guidelines from the Infectious Diseases Society of America. Clin Infect Dis. 2010 Mar 1;50(5):625-63. doi: 10.1086/650482. PMID 20175247
- [Background] Nie ZL, Zhang KQ, Li QS, Jin FS, Zhu FQ, Huo WQ. Treatment of urinary fistula after kidney transplantation. Transplant Proc. 2009 Jun;41(5):1624-6. doi: 10.1016/j.transproceed.2008.10.103. PMID 19545693
- [Background] Kumar A, Verma BS, Srivastava A, Bhandari M, Gupta A, Sharma R. Evaluation of the urological complications of living related renal transplantation at a single center during the last 10 years: impact of the Double-J* stent. J Urol. 2000 Sep;164(3 Pt 1):657-60. doi: 10.1097/00005392-200009010-00010. PMID 10953120
- [Background] Erbas B. Peri- and Postsurgical Evaluations of Renal Transplant. Semin Nucl Med. 2017 Nov;47(6):647-659. doi: 10.1053/j.semnuclmed.2017.07.002. Epub 2017 Jul 25. PMID 28969763
- [Background] Rigg KM, Proud G, Taylor RM. Urological complications following renal transplantation. A study of 1016 consecutive transplants from a single centre. Transpl Int. 1994;7(2):120-6. PMID 8179799
- [Background] Karam G, Hetet JF, Maillet F, Rigaud J, Hourmant M, Soulillou JP, Giral M. Late ureteral stenosis following renal transplantation: risk factors and impact on patient and graft survival. Am J Transplant. 2006 Feb;6(2):352-6. doi: 10.1111/j.1600-6143.2005.01181.x. PMID 16426320
- [Background] Golebiewska JE, Debska-Slizien A, Rutkowski B. Urinary tract infections during the first year after renal transplantation: one center's experience and a review of the literature. Clin Transplant. 2014 Nov;28(11):1263-70. doi: 10.1111/ctr.12465. Epub 2014 Oct 15. PMID 25251447
- [Background] Alberts VP, Idu MM, Legemate DA, Laguna Pes MP, Minnee RC. Ureterovesical anastomotic techniques for kidney transplantation: a systematic review and meta-analysis. Transpl Int. 2014 Jun;27(6):593-605. doi: 10.1111/tri.12301. Epub 2014 Apr 8. PMID 24606191
- [Background] Hollyer I, Ison MG. The challenge of urinary tract infections in renal transplant recipients. Transpl Infect Dis. 2018 Apr;20(2):e12828. doi: 10.1111/tid.12828. Epub 2018 Jan 25. PMID 29272071
- [Background] Lee JR, Bang H, Dadhania D, Hartono C, Aull MJ, Satlin M, August P, Suthanthiran M, Muthukumar T. Independent risk factors for urinary tract infection and for subsequent bacteremia or acute cellular rejection: a single-center report of 1166 kidney allograft recipients. Transplantation. 2013 Oct 27;96(8):732-8. doi: 10.1097/TP.0b013e3182a04997. PMID 23917724
- [Background] Shams SF, Eidgahi ES, Lotfi Z, Khaledi A, Shakeri S, Sheikhi M, Bahrami A. Urinary tract infections in kidney transplant recipients 1st year after transplantation. J Res Med Sci. 2017 Feb 16;22:20. doi: 10.4103/1735-1995.200274. eCollection 2017. PMID 28458711
- [Background] Mahdavi-Zafarghani R, Taghavi R. Urological complications following renal transplantation: assessment in 500 recipients. Transplant Proc. 2002 Sep;34(6):2109-10. doi: 10.1016/s0041-1345(02)02870-1. No abstract available. PMID 12270332